CLINICAL TRIAL: NCT01400126
Title: The Effect of Ultrapure Water System on Hemodialysis Therapy- a Single Center Trial
Brief Title: Ultrapure Water System for Hemodialysis Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Prof. Doron Schwartz, TelAvivMC
Other Study IDs: 01
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-11

CONDITIONS: The Change of Biomarkers CRP, CBC With the Use of Ultra Pure Water System for; Hemodialysis.; The Rate of Adverse Events Such as Hypotension During Hemodialysis Therapy With Ultra Pure Water; System as Compared to Conventional Water System.
Keywords: Ultrapure water,hemodialysis, CRP, blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We wish to compare the effect of very clean water used for dialysis therapy (i.e ultrapure water) in comparison with the use of conventional water which are used in most dialysis units worldwide. To the best of our knowledge prospective data in that field is sparse.

DETAILED DESCRIPTION:
In observational studies, the use of very pure dialysis solution has been suggested to reduce the plasma level of CRP, IL-6 ; to improve the response to anemia to erythropoietin therapy ; to promote better nutrition as evidenced by increase in plasma albumin value , estimated dry body weight, midarm muscle circumference and urea-nitrogen appearance rate; to reduce plasma level of β2-microglobulin and pentosidine ; to dely carpal tunnel syndrome ; to slow the loss of residual renal function; and to lower cardiovascular morbidity.The aim of this study is to prospectively evaluate the effect of dialysis performed with ultra-pure water (UPW)in comparison with dialysis with the use of conventional water system. Patients enrolled into this study will be evaluated at initial period of one month treated with conventional water system (-30 to 0 days). Then water system will be switched to ultra-pure water system with the use of filter added to the dialysis machine (Gambro). After switching to UPW system the patients will be followed for a period of one year (days 0-365). Primary end point will be change in CRP. Additional parameters: Blood pressure, adverse events during dialysis, hemoglobin levels and white-blood cell counts.

ELIGIBILITY:
Inclusion Criteria:

1. chronic hemodialysis therapy thrice weekly > 3 months of therapy
2. Signed an informed consent -

Exclusion Criteria:

1. Enrolled to other study
2. Ongoing infection -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
CRP | 13 months

SECONDARY OUTCOMES:
blood pressure | 13 months